CLINICAL TRIAL: NCT00627406
Title: A Prospective Randomised Study to Evaluate the Effect of Triggering Ovulation With GnRHa (Buserelin) and Low Dose hCG (Pregnyl) as Compared to the Use of Conventional Doses of hCG (Pregnyl)
Brief Title: Triggering of Final Oocyte Maturation With GnRHa (Buserelin) in GnRH Antagonist Cycles
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Regionshospitalet Viborg, Skive (Other)
Responsible Party: Principal Investigator, Peter Humaidan, Prof. M.D. D.M.Sc., Regionshospitalet Viborg, Skive
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: N-VN-2002-0046MCH
Record Dates: First submitted 2008-02-22; First posted 2008-03-03 (Estimated); Results first posted 2013-11-27 (Estimated); Last update posted 2013-11-27 (Estimated); Status verified 2013-09

CONDITIONS: OHSS (Ovarian Hyperstimulation)
Keywords: GnRH antagonist; GnRH agonist; hCG; OHSS; In vitro fertilization; ovulation induction; Clinical pregnancy rate
MeSH Terms: conditions — Ovarian Hyperstimulation Syndrome | interventions — Buserelin; Chorionic Gonadotropin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- A (Experimental): More than 14 follicles with a diameter of > 11mm: triggering of ovulation with 0.5 mg GnRHa (Buserelin) (s.c.) + 1500 IU hCG (Pregnyl)
  Interventions: Drug: Buserelin and Pregnyl
- B (Active Comparator): More than 14 follicles with a diameter of > 11mm: triggering of ovulation with hCG (Pregnyl) 5.000 IU (s.c.)
  Interventions: Drug: Pregnyl
- C (Experimental): 14 or less follicles with a diameter of > 11mm: triggering of ovulation with 0.5 mg GnRHa (Buserelin) (s.c.) + 1500 IU hCG (Pregnyl) (s.c.) at 35 hours and 1500 IU hCG (Pregnyl) (s.c.) 7 days after triggering of ovulation (OPU + 5)
  Interventions: Drug: Buserelin and Pregnyl
- D (Active Comparator): 14 or less follicles with a diameter of > 11mm: triggering of ovulation with 5000 IU hCG (Pregnyl) (s.c.)
  Interventions: Drug: Pregnyl

INTERVENTIONS:
Drug: Buserelin and Pregnyl — Subcutaneous injection 0.5 mg and 1500 IU
  Arms: A
Drug: Pregnyl — Subcutaneous injection 5000 IU
  Arms: B
Drug: Buserelin and Pregnyl — Subcutaneous injection 0,5 mg and 1500 IU + 1500 IU after 7 days
  Arms: C
Drug: Pregnyl — Subcutaneous injection 5000 IU
  Arms: D

SUMMARY:
The purpose of this study is to possibly further improve the clinical outcome and explore the incidence of OHSS in patients, who have final oocyte maturation with GnRHa (Buserelin) in GnRH antagonist IVF/ICSI cycles

ELIGIBILITY:
Inclusion Criteria:

* Patient complying with the conditions for IVF or ICSI treatment
* Female age over 20 years and under 40 years
* Normal regular cycle and patients with oligomenorrhea
* BMI > 18 and < 35
* each patient contributes with one cycle only

Exclusion Criteria:

* Significant disturbances in the woman (diabetes, epilepsy, liver/renal/heart disease, metabolic disorder)
* Patients with > 25 follicles on the day of triggering ovulation

Ages: 20 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 384 (Actual)
Dates: Start 2009-01; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter S Humaidan, MD, Principal Investigator
Locations (1):
- The Fertility Clinic, Regional Hospital of Skive, Skive, Denmark

REFERENCES:
- [Derived] Humaidan P, Polyzos NP, Alsbjerg B, Erb K, Mikkelsen AL, Elbaek HO, Papanikolaou EG, Andersen CY. GnRHa trigger and individualized luteal phase hCG support according to ovarian response to stimulation: two prospective randomized controlled multi-centre studies in IVF patients. Hum Reprod. 2013 Sep;28(9):2511-21. doi: 10.1093/humrep/det249. Epub 2013 Jun 9. PMID 23753114

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period from jan. 2009 to dec. 2011. Participanting Clinics Fertility clinic Regional Hospital Skive, University Hostipal Odense, Regional Hospital Holbaek, Denmark.
Groups:
- A: >14 Follicles; GnRHa Trigger + 1500 hCG: More than 14 follicles with a diameter of > 11mm: triggering of ovulation with 0.5 mg GnRHa (Buserelin) (s.c.) + 1500 IU hCG (Pregnyl)
  Buserelin and Pregnyl : Subcutaneous injection 0.5 mg and 1500 IU
- B: >14 Follicles; hCG Trigger: More than 14 follicles with a diameter of > 11mm: triggering of ovulation with hCG (Pregnyl) 5.000 IU (s.c.)
  Pregnyl : Subcutaneous injection 5000 IU
- C:<15 Follicles; GnRHa Trigger + 1500 hCG x 2: 14 or less follicles with a diameter of > 11mm: triggering of ovulation with 0.5 mg GnRHa (Buserelin) (s.c.) + 1500 IU hCG (Pregnyl) (s.c.) at 35 hours and 1500 IU hCG (Pregnyl) (s.c.) 7 days after triggering of ovulation (OPU + 5)
  Buserelin and Pregnyl : Subcutaneous injection 0,5 mg and 1500 IU + 1500 IU after 7 days
- D: <15 Follicles; hCG Trigger: 14 or less follicles with a diameter of > 11mm: triggering of ovulation with 5000 IU hCG (Pregnyl) (s.c.)
  Pregnyl : Subcutaneous injection 5000 IU
Period: Overall Study
Arm/Group | A: >14 Follicles; GnRHa Trigger + 1500 hCG | B: >14 Follicles; hCG Trigger | C:<15 Follicles; GnRHa Trigger + 1500 hCG x 2 | D: <15 Follicles; hCG Trigger
Started | 60 | 58 | 125 | 141
Completed | 60 | 58 | 125 | 141
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | A: >14 Follicles; GnRHa Trigger + 1500 hCG | B: >14 Follicles; hCG Trigger | C:<15 Follicles; GnRHa Trigger + 1500 hCG x 2 | D: <15 Follicles; hCG Trigger | Total
Number analyzed (Participants) | 60 | 58 | 125 | 141 | 384
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 60 | 58 | 125 | 141 | 384
  >=65 years | 0 | 0 | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 28.5 (5.2) | 29.8 (3.8) | 30.8 (3.9) | 31.5 (3.7) | 30.2 (4.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60 | 58 | 125 | 141 | 384
  Male | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Denmark | 60 | 58 | 125 | 141 | 384

OUTCOME MEASURES:

1. Primary Outcome: Frequency of Moderate to Severe OHSS.
Time Frame: From the date of triggering ovulation until 2 weeks after pregnancy test. group C and D. 12 days after pregnancy test
Population: No power calculation was proformed.
Measure: Number; unit: participants
Arm/Group | A: >14 Follicles; GnRHa Trigger + 1500 hCG | B: >14 Follicles; hCG Trigger | C:<15 Follicles; GnRHa Trigger + 1500 hCG x 2 | D: <15 Follicles; hCG Trigger
Number analyzed (Participants) | 60 | 58 | 125 | 141
participants | 0 | 2 | 2 | 0

2. Secondary Outcome: Pregnancy Rate
Time Frame: from stimulation day 1 until last ultrasound scan 7 weeks after a positive pregnancy test
Measure: Number; unit: participants
Arm/Group | A: >14 Follicles; GnRHa Trigger + 1500 hCG | B: >14 Follicles; hCG Trigger | C:<15 Follicles; GnRHa Trigger + 1500 hCG x 2 | D: <15 Follicles; hCG Trigger
Number analyzed (Participants) | 60 | 58 | 125 | 141
participants | 17 | 15 | 37 | 36

ADVERSE EVENTS:
Arm/Group | A: >14 Follicles; GnRHa Trigger + 1500 hCG | B: >14 Follicles; hCG Trigger | C:<15 Follicles; GnRHa Trigger + 1500 hCG x 2 | D: <15 Follicles; hCG Trigger
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/58 | 0/125 | 0/141
Other Adverse Events (participants affected / at risk) | 0/60 | 0/58 | 0/125 | 0/141

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No